CLINICAL TRIAL: NCT03698097
Title: Patient Surveys - What Patients Want
Acronym: ch18Saxer
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-01845; ch18Saxer
Record Dates: First submitted 2018-10-04; First posted 2018-10-05 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Patient Survey
Keywords: quality management; paper questionnaires; satisfaction surveys; survey technique; online questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: patient satisfaction survey — Patient survey completed in a paper or survey monkey based internet version accessible via a QR code or link

SUMMARY:
This study is to gain insight into patients' preferences considering satisfaction surveys, specifically asking for their most pressing topics and their preferred survey technique.

DETAILED DESCRIPTION:
The practice of patient surveys for quality management is revised at the University Hospital Basel (USB). One aspect is a more versatile data acquisition via online portals and/or paper questionnaires, another aspect is the content of questions and the assessment of demographic data. In this situation a tentative survey on their preferences in this context was realised in patients who were treated in autumn 2016 at the Department of Orthopaedics and Trauma Surgery (DOTS) using a cover letter informing them about the nature of the survey. They were asked to provide few basic demographic data, they were furthermore asked whether they favoured surveys by the USB and if so with which focus. Finally they had the option to name three central topics for feedback and to quantify the number of questionnaires they had so far received by the USB. The survey could be completed in a paper and survey monkey based internet version accessible via a Quick Response (QR) code or link.

ELIGIBILITY:
Inclusion Criteria:

* All data from completed survey sheets (paper questionnaires) and online forms are included

Exclusion Criteria:

* no exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Data were collected from a random sample of patients after out- or inpatient treatment at the DOTS
Sampling Method: Probability Sample
Enrollment: 745 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
patients' preferences considering preferred survey technique | after out- or inpatient treatment at the DOTS in a three months period in autumn 2016
  patients' preferences considering paper questionnaire or survey monkey based internet version accessible via a QR code or link

SECONDARY OUTCOMES:
patients' preferences asking for their most pressing topics | after out- or inpatient treatment at the DOTS in a three months period in autumn 2016
  option to name three central topics for feedback

CONTACTS AND LOCATIONS:
Overall Officials: Franziska Saxer, Dr. med, Principal Investigator — Department of Orthopaedics and Trauma Surgery (DOTS).
Locations (1):
- Department of Orthopaedics and Trauma Surgery (DOTS)., Basel, Switzerland